CLINICAL TRIAL: NCT02778074
Title: Internet-guided Cognitive Behavioural Therapy to Improve Depression in Patients With Cardiovascular Disease
Brief Title: Internet-guided Cognitive Behavioural Therapy to Improve Depression Patients With Cardiovascular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Peter Johansson, RN, PhD, Professor, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-02600
Record Dates: First submitted 2016-05-16; First posted 2016-05-19 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-11

CONDITIONS: Cardiovascular Disease; Depression
Keywords: Internet Cognitive Behavioural Therapy
MeSH Terms: conditions — Cardiovascular Diseases; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet Cognitive Behavioural Therapy (Experimental): Participants will perform a nine-week tailored I-CBT program developed to fit CVD patients. The program consists of psychoeducation, relaxation, problem-solving and behavioral activation.
  Interventions: Behavioral: Internet cognitive behavioural therapy
- Moderated discussion forum (Placebo Comparator): In this arm the participants are allocated to a non mandatory discussion forum for nine weeks. Evert week will participants discuss issues regarding their CVD. Themes discussed are suggested by the study team, and a new theme is added every week. A moderator from the study group act as a supervisor and checks that issues discussed are ok. After the nine week discussion forum the participants are offered the nine week CBT program.
  Interventions: Behavioral: Moderated Discussion Forum

INTERVENTIONS:
Behavioral: Internet cognitive behavioural therapy — A nine-week tailored I-CBT program for patients with CVD. The CBT program consists of the components of psychoeducation, relaxation, problem-solving and behavioural activation.
  Other Names: I-CBT
  Arms: Internet Cognitive Behavioural Therapy
Behavioral: Moderated Discussion Forum — Participants will be allocated to an internet moderated discussion forum during 9 weeks. Patients will discuss issues related to cardiovascular disease. A new topic will be discussed every week. After 9 weeks, those in the moderated discussion forum will be offered to perform the I-CBT program.
  Arms: Moderated discussion forum

SUMMARY:
Purpose and aims Tailored internet-based cognitive behavioural therapy (I-CBT) is a new innovative and person-centred method that is promising that may be used to decrease depression in patients with cardiovascular disease (CVD). In patients with CVD, depressive symptoms is a common co-morbidity leading to decreased wellbeing, and increased morbidity and mortality. Depressive symptoms are both underdiagnosed and undertreated in CVD patients. Earlier studies have demonstrated the efficiency of cognitive behavioural therapy (CBT) for many psychiatric conditions, but few studies have evaluated CBT in patients with CVD.

The overall purpose of this study is to evaluate the effects of the tailored I-CBT program on reducing depressive symptoms and other patient reported outcomes in patients with cardiovascular disease (CVD) and to explore factors related to implementation of the I-CBT program in clinical cardiac care.

The primary aim:

-To evaluate the effects of the tailored I-CBT depression program on depressive symptoms.

Secondary aims:

* To evaluate effects on quality of life´, sleep and anxiety
* To evaluate factors that can influence the I-CBT programs effect on depressive symptoms.
* To gain knowledge about the I-CBT program, as perceived by patients and health care professionals.
* To explore facilitators and barriers to the implementation of the I-CBT program in clinical practice from the perspectives of patients, health care professionals and policymakers.

DETAILED DESCRIPTION:
Power calculation: Effect size=0.5, alpha=0.05 (Z=1.96), Power 0.80 (Z -0.84) = 122 participants. Due to drop-outs or deaths the size of the study population for the RCT study was decided to n=140.

ELIGIBILITY:
Inclusion Criteria:

* treatment for CVD according to European Society of Cardiology guidelines.
* stable CVD (NYHA class I-III) and not having been hospitalised for CVD in in the last four weeks.
* depressive symptoms (Patient Health Questionnaire-9 17 (PHQ-9) > 5 points)

Exclusion Criteria:

* severe CVD (NYHA IV) or another severe chronic life-threatening disease
* severe depression assessed as requiring acute treatment
* not being able to dedicate 3-4 hours to participate in the program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Johansson, PhD, Principal Investigator — Department of Social and Welfare Studies, Linköping University, Norrköping, Sweden
Locations (1):
- Linkoping University, Norrköping, Sweden

REFERENCES:
- [Derived] Mourad G, Lundgren J, Andersson G, Johansson P. Healthcare use in patients with cardiovascular disease and depressive symptoms - The impact of a nurse-led internet-delivered cognitive behavioural therapy program. A secondary analysis of a RCT. Internet Interv. 2023 Dec 5;35:100696. doi: 10.1016/j.invent.2023.100696. eCollection 2024 Mar. PMID 38093803
- [Derived] Westas M, Mourad G, Andersson G, Lundgren J, Johansson P. The effects of internet-based cognitive behaviour therapy for depression in cardiovascular disease on symptoms of anxiety: a secondary analysis of a randomized trial. Eur J Cardiovasc Nurs. 2024 May 28;23(4):382-390. doi: 10.1093/eurjcn/zvad097. PMID 37740442
- [Derived] Johansson P, Lundgren J, Andersson G, Svensson E, Mourad G. Internet-Based Cognitive Behavioral Therapy and its Association With Self-efficacy, Depressive Symptoms, and Physical Activity: Secondary Analysis of a Randomized Controlled Trial in Patients With Cardiovascular Disease. JMIR Cardio. 2022 Jun 3;6(1):e29926. doi: 10.2196/29926. PMID 35657674
- [Derived] Mourad G, Lundgren J, Andersson G, Husberg M, Johansson P. Cost-effectiveness of internet-delivered cognitive behavioural therapy in patients with cardiovascular disease and depressive symptoms: secondary analysis of an RCT. BMJ Open. 2022 Apr 11;12(4):e059939. doi: 10.1136/bmjopen-2021-059939. PMID 35410939
- [Derived] Westas M, Lundgren J, Andersson G, Mourad G, Johansson P. Effects of Internet-delivered cognitive behavioural therapy adapted for patients with cardiovascular disease and depression: a long-term follow-up of a randomized controlled trial at 6 and 12 months posttreatment. Eur J Cardiovasc Nurs. 2022 Aug 29;21(6):559-567. doi: 10.1093/eurjcn/zvab131. PMID 35061868
- [Derived] Johansson P, Westas M, Andersson G, Alehagen U, Brostrom A, Jaarsma T, Mourad G, Lundgren J. An Internet-Based Cognitive Behavioral Therapy Program Adapted to Patients With Cardiovascular Disease and Depression: Randomized Controlled Trial. JMIR Ment Health. 2019 Oct 3;6(10):e14648. doi: 10.2196/14648. PMID 31584000

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Internet Cognitive Behavioural Therapy | Moderated Discussion Forum
Started | 72 | 72
Completed | 65 | 62
Not Completed | 7 | 10
Not completed — Lost to Follow-up | 7 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Internet Cognitive Behavioural Therapy | Moderated Discussion Forum | Total
Number analyzed (Participants) | 72 | 72 | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (13) | 64 (12) | 63 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Gender: Female | 25 | 30 | 55
  Gender: Male | 47 | 42 | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 72 | 72 | 144
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 72 | 72 | 144
Depression by Patient Health Questonnaire-9 (range 0-27, higher numbers represents more depression [Mean (Standard Deviation); unit: units on a scale] | 10.71 (4.47) | 10.22 (5.10) | 10.47 (4.78)

OUTCOME MEASURES:

1. Primary Outcome: Depressive Symptoms Collected With the Patient Health Questionnaire-9 (PHQ-9)
Description: The PHQ-9 is a nine-item instrument for measurement of depressive symptoms during the last two weeks. Each item is answered on a four graded scale where zero represents that the item do not affect the person and numbers one to three represents that the item affects the person several days to almost every day. The answers are summed to a total sum score, range 0-27, with higher numbers representing higher level of depressive symptoms. A cut off >5 represents minor depression and a cut off >10 represents major depression
Time Frame: Score at 9 weeks follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Internet Cognitive Behavioural Therapy | Moderated Discussion Forum
Number analyzed (Participants) | 72 | 72
score on a scale | 6.63 (4.76) | 8.68 (4.60)
Statistical Analysis 1: Comparison: Internet Cognitive Behavioural Therapy vs Moderated Discussion Forum; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = -2.34

ADVERSE EVENTS:
Time Frame: 9 weeks
Arm/Group | Internet Cognitive Behavioural Therapy | Moderated Discussion Forum
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/72
Other Adverse Events (participants affected / at risk) | 0/72 | 0/72

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-28): https://cdn.clinicaltrials.gov/large-docs/74/NCT02778074/Prot_SAP_001.pdf